CLINICAL TRIAL: NCT04633122
Title: A Multicenter Phase 2, Single-Arm Open-Label Study of DCC-2618 to Assess Efficacy, Safety, and Pharmacokinetics In Patients With Advanced Gastrointestinal Stromal Tumors Who Have Progressed On Prior Anticancer Therapies
Brief Title: A Study to Assess DCC-2618 and Sunitinib in Patients With Advanced GIST After Treatment With Imatinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZL-2307-003
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Stromal Tumor(GIST)
Keywords: Gastrointestinal Stromal Tumors,GIST,DCC-2618,Ripretinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ripretinib (Experimental): 50mg/tablet,150 mg QD continuous administration, 6 weeks (42 days) for a cycle.
  Interventions: Drug: Ripretinib
- Sunitinib (Active Comparator): 12.5mg/capsule, 50 mg QD, in 6 weeks (42 days) with 4 weeks continuous dosing followed by 2 weeks break.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Ripretinib — Oral kinase inhibitor
  Other Names: DCC-2618
  Arms: Ripretinib
Drug: Sunitinib — second-line therapy in GIST patients who have progressed after imatinib treatment or are intolerant to imatinib
  Arms: Sunitinib

SUMMARY:
the primary objective of this study is to assess the efficacy (progression-free survival,PFS) of DCC-2618 (ripretinib, ZL-2307) and sunitinib in patients with advanced gastrointestinal stromal tumors after treatment with imatinib. This study will enroll approximately 98 subjects in around 18 sites in China mainland, and all subjects will be receiving DCC-2618 or Sunitinib in equal chance as treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age.
* Histological diagnosis of advanced GIST and capability of providing tumor tissue sample (the interval between tumor tissue collection and signing of informed consent form should be less than 3 years). Otherwise, biopsy is required.
* Provide molecular test report with KIT/PDGFRA mutation status prior to randomization.
* Patients must have progressed on imatinib or have documented intolerance to imatinib. Subjects must have discontinued imatinib treatment 10 days prior to the first dose of the study drug. All prior imatinib treatments will be considered as first-line (such as imatinib adjuvant therapy and imatinib dose increase).
* ECOG PS of 0-2.
* Female patients of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at screening.
* Patients of reproductive potential must agree to follow the contraception requirements.
* At least 1 measurable lesion according to the "RECIST v1.1-GIST-specific Criteria" (non-nodal lesions must be ≥1.0 cm in the long axis or ≥ double the slide thickness in the long axis) ; obtaining radiographic image results within 28 days prior to the first dose of study drug.
* Good organ function and bone marrow reserve function, including:

  * Neutrophil count ≥ 1,000/µL
  * Hemoglobin ≥ 8 g/dL
  * Platelet count ≥ 75,000/µL
  * Total bilirubin ≤ 1.5 × the upper limit of normal (ULN)
  * AST and ALT ≤ 3×ULN, and AST and ALT≤ 5×ULN in the presence of hepatic metastases
  * Creatinine clearance ≥ 50 mL/min (based on Cockcroft-Gault estimation Formulas for calculation)
  * Prothrombin time (PT), international normalized ratio (INR) or partial thromboplastin time ≤ 1.5 × ULN. Patients on a stable, maintenance regimen of anticoagulant therapy for at least 30 days prior to study drug administration may have PT/INR measurements >1.5 × ULN if, in the opinion of the investigator, the patient is suitable for the study. An adequate rationale must be provided to the sponsor prior to randomization.
* Resolution of all toxicities from prior therapy to ≤Grade 1 (or baseline) within 1 week prior to the first dose of study drug (excluding alopecia and ≤ Grade 3 clinically asymptomatic lipase, amylase, and creatine phosphokinase laboratory abnormalities).
* Patient is capable of understanding and complying with the protocol. Subjects should sign the written informed consent before any study-related procedures were performed.

Exclusion Criteria:

* Treatment with any other line of therapy in addition to imatinib for advanced GIST. Imatinib-containing combination therapy in the first-line treatment should not be enrolled.
* Patients with a prior or concurrent malignancy whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of this clinical trial are not eligible.
* Patient has known active central nervous system metastases.
* New York Heart Association class II - IV heart disease, myocardial infarct, active ischemia or any other uncontrolled cardiac condition within the first 6 months of the first dose of study drug such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension or congestive heart failure.
* Left ventricular ejection fraction (LVEF) < 50%.
* Arterial thrombotic or embolic events such as cerebrovascular accident (including ischemic attacks) or hemoptysis within 6 months before the first dose of study drug.
* Venous thrombotic events (e.g. deep vein thrombosis) or pulmonary arterial events (e.g. pulmonary embolism) within 1 month before the first dose of study drug. Patients on stable anticoagulation therapy for at least one month are eligible.
* 12-lead electrocardiogram (ECG) demonstrating QT interval corrected by Fridericia's formula > 450 ms in males or > 470 ms in females at screening or history of long QT interval syndrome.
* Use of strong or moderate inhibitors and/or inducers of cytochrome P450 (CYP) 3A4 within 14 days or 5 x the half-life (whichever is longer) prior to the first dose of study drug, including certain herbal medications (eg, St. John's Wort) and consumption of grapefruit or grapefruit juice within 14 days prior to the first dose of study drug.
* Use of known substrates or inhibitors of breast cancer resistance protein (BCRP) transporters within 14 days or 5 x the half-life (whichever is longer) prior to the first dose of study drug.
* Major surgeries (e.g. abdominal laparotomy) within 4 weeks of the first dose of study drug; all major surgical wounds must be healed and free of infection or dehiscence before the first dose of study drug.
* Any other clinically significant comorbidities, such as uncontrolled pulmonary disease, active infection, or any other condition, which in the judgment of the investigator, could compromise compliance with the protocol, interfere with interpretation of the study results, or predispose the patient to safety risks.
* Known human immunodeficiency virus or hepatitis C infection only if the patient is taking medications that are excluded per protocol, hepatitis B virus (HBV) DNA > 2000 IU/ml or > 104 copies/ml.
* Female patients who are pregnant or lactating or who plan to become pregnant during the study treatment period.
* Known hypersensitivity to any component of the study drug. Patients with Stevenson Johnson syndrome in previous TKI treatment need to be excluded.
* Gastrointestinal abnormalities including but not limited to:

  * inability to take oral medication
  * malabsorption syndrome
  * Requiring intravenous nutrition
* Any active hemorrhages, excluding hemorrhoids or gum bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The General Hospital of Peking University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical Universty, Chongqing, Chognqing
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The Cancer Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The sixth Affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The 4th Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Affiliated Hospital of Haerbin MedicalUniversity, Harbin, Heilongjiang
  - Union Hospital of HUST, Wuhan, Hubei
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Fudan University, Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 108 patients were randomized.
Period: Overall Study
Arm/Group | Ripretinib | Sunitinib
Started | 54 | 54
Completed | 13 | 15
Not Completed | 41 | 39
Not completed — Remained on treatment | 19 | 14
Not completed — Survival follow-up stopped | 22 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ripretinib | Sunitinib | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 39 | 74
  >=65 years | 19 | 15 | 34
Age, Continuous [Median (Full Range); unit: years] | 59 [25 to 82] | 58.5 [28 to 81] | 59 [25 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 36 | 33 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 54 | 54 | 108
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time interval from randomization to the first occurrence of progressive disease based on assessment of the independent radiology review (IRR) or death due to any causes.
Time Frame: Approximately 12 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ripretinib | Sunitinib
Number analyzed (Participants) | 54 | 54
months | 10.3 [5.5 to NA] — The upper limit of 95% CI was not evaluable due to low PFS maturity. | 8.3 [4.9 to NA] — The upper limit of 95% CI was not evaluable due to low PFS maturity.

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The percentage of participants whose efficacy is confirmed as complete response (CR) or partial responses (PR) based on independent radiology review.
Time Frame: Approximately 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Ripretinib | Sunitinib
Number analyzed (Participants) | 54 | 54
Participants | 16 | 11

3. Secondary Outcome: Disease Control Rate (DCR)
Description: The percentage of participants whose efficacy is confirmed as complete response (CR) or partial responses (PR) or duration of SD ≥ 12 months based on independent radiology review.
Time Frame: Approximately 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Ripretinib | Sunitinib
Number analyzed (Participants) | 54 | 54
Participants | 24 | 20

ADVERSE EVENTS:
Time Frame: Approximately 12 months.
Description: An AE is defined as any untoward medical occurrence in a patient administered a pharmaceutical product during the study, which does not necessarily have a causal relationship with the study drug. This includes any newly occurring event or previous condition that has increased in severity or frequency after the ICF is signed.
Arm/Group | Ripretinib | Sunitinib
All-Cause Mortality (participants affected / at risk) | 13/54 | 15/54
Serious Adverse Events (participants affected / at risk) | 9/54 | 12/54
Other Adverse Events (participants affected / at risk) | 54/54 | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ripretinib (N=54) | Sunitinib (N=54)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ripretinib (N=54) | Sunitinib (N=54)
Alopecias (Skin and subcutaneous tissue disorders) | 27 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 4
Anaemia (Blood and lymphatic system disorders) | 17 | 40
Hypothyroidism (Endocrine disorders) | 10 | 17
Abdominal pain (Gastrointestinal disorders) | 16 | 10
Asthenia (General disorders) | 15 | 10
Blood bilirubin increased (Investigations) | 17 | 19
Weight decreased (Investigations) | 17 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 15
Neutrophil count decreased (Investigations) | 1 | 42
White blood cell count decreased (Investigations) | 1 | 41
Platelet count decreased (Investigations) | 3 | 34
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 7
Constipation (Gastrointestinal disorders) | 11 | 4
Diarrhoea (Gastrointestinal disorders) | 11 | 13
Blood creatine phosphokinase increased (Investigations) | 5 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 11
Hypertesion (Vascular disorders) | 16 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 | 29
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 16
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Proteinuria (Renal and urinary disorders) | 8 | 6
Headache (Nervous system disorders) | 6 | 4
Dizziness (Nervous system disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 4
Hypoproteinaemia (Metabolism and nutrition disorders) | 4 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8 | 6
Lymphocyte count decreased (Investigations) | 2 | 8
Aspartate aminotransferase increased (Investigations) | 3 | 13
Alanine aminotransferase increased (Investigations) | 4 | 8
Influenza like illness (General disorders) | 5 | 1
Pyrexia (General disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 3 | 7
Flatulence (Gastrointestinal disorders) | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 4
Sinus arrhythmia (Cardiac disorders) | 1 | 3
Sinus bradycardia (Cardiac disorders) | 3 | 1
Periorbital swelling (Eye disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 9 | 3
Gingival bleeding (Gastrointestinal disorders) | 7 | 2
Nausea (Gastrointestinal disorders) | 5 | 3
Toothache (Gastrointestinal disorders) | 6 | 3
Chest discomfort (General disorders) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 4
Urinary tract infection (Infections and infestations) | 4 | 1
Bilirubin conjugated increased (Investigations) | 5 | 3
Blood bilirubin unconjugated increased (Investigations) | 4 | 4
Blood creatinine increased (Investigations) | 4 | 4
Blood lactate dehydrogenase increased (Investigations) | 4 | 7
Blood thyroid stimulating hormone increased (Investigations) | 0 | 7
High density lipoprotein decreased (Investigations) | 3 | 3
Lipase increased (Investigations) | 4 | 3
Neutrophil count increased (Investigations) | 7 | 2
Occult blood positive (Investigations) | 0 | 3
Prealbumin decreased (Investigations) | 3 | 3
White blood cell count increased (Investigations) | 8 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Insomnia (Psychiatric disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT04633122/Prot_SAP_000.pdf